CLINICAL TRIAL: NCT02553395
Title: One Week Assessment of The Phenacite Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CV-15-40
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenacite contact lens (Experimental): Study Test Contact Lens
  Interventions: Device: Phenacite (Test) contact lens
- comfilcon A contact lens (Active Comparator): Control Contact Lens
  Interventions: Device: comfilcon A contact lens

INTERVENTIONS:
Device: Phenacite (Test) contact lens
  Arms: Phenacite contact lens
Device: comfilcon A contact lens
  Arms: comfilcon A contact lens

SUMMARY:
This study will investigate performance criteria over one week of daily wear to determine if the Study Test contact lens performs equivalently to the comfilcon A contact lenses in terms of subjective ratings and of visual performance.

The study test lens was not the final optical design and the study results were not used for the design validation.

DETAILED DESCRIPTION:
This will be double-masked, randomized, bilateral crossover study comparing the Study Test lens against the comfilcon A control lens, each worn over one week of daily wear.

The study test lens was not the final optical design and the study results were not used for the design validation.

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if he/she:

  * Oculo-visual examination in the last two years
  * Between 18 and 35 years of age and has full legal capacity to volunteer
  * Has read and understood the informed consent letter
  * Is willing and able to follow instructions and maintain the appointment schedule
  * Is correctable to a visual acuity of 20/25 or better (in each eye) with their habitual correction or 20/20 best corrected
  * Currently wears, or has previously successfully worn, soft contact lenses between -1.00D (Diopter) and -4.50D
  * Spherical Contact Lens Rx between -1.00 and -4.00 and spectacle cylinder <-0.75
  * Currently spends a minimum of 4 hours a day; 5 days a week on digital devices and can replicate this time during the study period
  * Is willing and able to wear the study contact lenses a minimum of 10 hours per day; 5 days a week.

Exclusion Criteria:

* A person will be excluded from the study if he/she:

  * Has never worn contact lenses before.
  * Has any systemic disease affecting ocular health.
  * Is using any systemic or topical medications that will affect ocular health.
  * Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
  * Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
  * Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
  * Is aphakic.
  * Has undergone corneal refractive surgery.
  * Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kollbaum, OD, PhD, Principal Investigator — Clinical Optics Research Lab (CORL)
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenacite Contact Lens Then Comfilcon A: Subjects were randomized to wear test lenses for one week and then cross-over to comfilcon A contact lens for one week.
  Phenacite : Contact Lens comfilcon A: contact lens
- Comfilcon A Contact Lens Then Phenacite Contact Lens: Subjects were randomized to wear comfilcon A lenses for one week and then cross-over to test contact lens for one week.
  comfilcon A: contact lens Phenacite : Contact Lens
Period: First Intervention
Arm/Group | Phenacite Contact Lens Then Comfilcon A | Comfilcon A Contact Lens Then Phenacite Contact Lens
Started | 12 | 18
Completed | 12 | 18
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Phenacite Contact Lens Then Comfilcon A | Comfilcon A Contact Lens Then Phenacite Contact Lens
Started | 12 | 18
Completed | 12 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear test lens for one week and then cross-over to control lens for one week.
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Visual Acuity (VA) - High Illumination High Contrast
Description: Binocular Distance visual acuity High Illumination High Contrast was assessed using logMAR (0.02 logMAR= 1 letter)
Time Frame: Baseline - After 5 minutes of lens settling
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Phenacite Contact Lens: Subjects were randomized to wear test contact lens for one week.
  Phenacite: Contact lens
- Comfilcon A Contact Lens: Subjects were randomized to wear control contact lens for one week.
  comfilcon A: contact lens
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
logMAR | -0.22 (0.05) | -0.24 (0.05)

2. Primary Outcome: Binocular Distance Visual Acuity (VA) -High Illumination High Contrast
Description: Binocular Distance visual acuity High Illumination High Contrast was assessed using logMAR (0.02 logMAR= 1 letter)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
logMAR | -0.20 (0.05) | -0.22 (0.06)

3. Primary Outcome: Binocular Near Visual Acuity (VA) - High Illumination High Contrast
Description: Binocular Near Visual Acuity High Illumination High Contrast was assessed on logMAR VA (0.02 logMAR= 1 letter)
Time Frame: Baseline - after 5 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
logMAR | -0.18 (0.06) | -0.19 (0.07)

4. Primary Outcome: Binocular Near Visual Acuity (VA) - High Illumination High Contrast
Description: Binocular Near Visual Acuity High Illumination High Contrast was assessed on logMAR VA (0.02 logMAR= 1 letter)
Time Frame: 1-week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
logMAR | -0.19 (0.06) | -0.19 (0.06)

5. Primary Outcome: Binocular Distance Visual Acuity (VA) - Low Illumination High Contrast
Description: Binocular Distance Visual Acuity (VA) - Low Illumination High Contrast was assessed using logMAR VA (0.02 logMAR= 1 letter)
Time Frame: Baseline (After 5 minutes of lens settling)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
LogMAR | -0.02 (0.05) | -0.04 (0.07)

6. Primary Outcome: Binocular Distance Visual Acuity (VA) - Low Illumination High Contrast
Description: as for outcome 5
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
LogMAR | 0.00 (0.08) | -0.04 (0.06)

7. Primary Outcome: Binocular Near Visual Acuity (VA) - Low Illumination High Contrast
Description: Binocular Near Visual Acuity (VA) - Low Illumination High Contrast was assessed using logMAR VA (0.02 logMAR= 1 letter)
Time Frame: Baseline (after 5 minutes of lens settling)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
LogMAR | -0.00 (0.07) | 0.00 (0.07)

8. Primary Outcome: Binocular Near Visual Acuity (VA) - Low Illumination High Contrast
Description: Binocular Near Visual Acuity (VA) - Low Illumination High Contrast was assessed using logMAR VA (0.02 logMAR= 1 letter)
Time Frame: 1week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
LogMAR | -0.01 (0.08) | -0.00 (0.06)

9. Primary Outcome: Subjective Ratings for Distance Quality of Vision
Description: Patient subjective scoring using anchors on the scale to provide a score between 0-100 for Distance Quality of Vision: (0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 30
score on a scale
  Phenacite Test Contact Lens | 85 (15)
  comfilcon A control lens | 91 (9)

10. Primary Outcome: Subjective Ratings for Intermediate Quality of Vision
Description: Patient subjective scoring using anchors on the scale to provide a score between 0-100 for Intermediate Quality of Vision: (0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 30
score on a scale
  Phenacite Test Lens | 91 (10)
  comfilcon A control lens | 95 (7)

11. Primary Outcome: Subjective Ratings for Near Quality of Vision
Description: Patient subjective scoring using anchors on the scale to provide a score between 0-100 for Near Quality of Vision: (0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 30
score on a scale
  Phenacite Test Lens | 92 (11)
  comfilcon A control lens | 95 (6)

12. Secondary Outcome: Post Blink Movement -
Description: Post blink movement was assessed by the investigator by the amount of movement (to the nearest 0.1mm) immediately after the blink (0.1mm steps)
Time Frame: Baseline (After 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
mm
  Right eye | 0.23 (0.06) | 0.24 (0.08)
  Left eye | 0.23 (0.06) | 0.25 (0.08)

13. Secondary Outcome: Post Blink Movement
Description: Investigator assessment of Amount of movement (to the nearest 0.1mm) immediately after the blink (0.1mm steps)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
mm
  Right eye | 0.24 (0.06) | 0.24 (0.07)
  Left Eye | 0.25 (0.08) | 0.25 (0.06)

14. Secondary Outcome: Push - Up Test for Lens Tightness
Description: Investigator assessment using Continuous Scale 0-100% (1% steps): 0%=Falls from cornea without lid support, 50%=Optimum, 100%=No movement
Time Frame: Baseline (After 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right eye | 50.83 (4.17) | 49.67 (2.92)
  Left Eye | 50.33 (4.14) | 49.17 (3.49)

15. Secondary Outcome: Push - Up Test for Lens Tightness
Description: as for outcome 14
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right Eye | 50.33 (4.14) | 49.17 (3.73)
  Left eye | 49.33 (6.53) | 49.17 (2.65)

16. Secondary Outcome: Lens Mobility Rating
Description: Investigator assessment using 5 Categories in 0.50 steps: 0=Immobile - no lag in any versions, 1=Restricted - no lag in some directions but slight lag (0-0.25mm) in others, 2=Secure - slight lag (0.25-0.5mm in each version), 3=Unrestricted - freely lags in a controlled manner on all versions, but not excessive (0.5-1.0mm), 4=Very mobile - excessive lag (>1mm) on versions in all directions in 0.25 steps
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right eye | 2.97 (0.20) | 3.00 (0.26)
  Left eye | 2.97 (0.22) | 3.02 (0.25)

17. Secondary Outcome: Lens Mobility Rating
Description: as for outcome 16
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right Eye | 2.98 (0.25) | 3.04 (0.16)
  Left eye | 3.02 (0.31) | 3.04 (0.16)

18. Secondary Outcome: Overall Lens Fit Acceptance
Description: Investigator assessment using 5 Categories in 0.25 steps: 0=Can't be worn, 1=Poor - should not be dispensed although no immediate danger, 2=Fair, 3=Good, 4=Optimum in 0.25 steps
Time Frame: Baseline (After 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right Eye | 3.48 (0.22) | 3.42 (0.36)
  Left Eye | 3.46 (0.22) | 3.44 (0.33)

19. Secondary Outcome: Overall Lens Fit Acceptance
Description: Investigator assessment using 5 Categories in 0.25 steps: 0=Can't be worn,, 1=Poor - should not be dispensed although no immediate danger, 2=Fair, 3=Good, 4=Optimum in 0.25 steps
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 30 | 30
units on a scale
  Right eye | 3.42 (0.28) | 3.48 (0.28)
  Left Eye | 3.35 (0.52) | 3.49 (0.28)

20. Secondary Outcome: Subjective Lens Preference - Distance Vision
Description: Patient subjective preference: Phenacite lens, comfilcon A or No Preference
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 30
percentage of participants
  Phenacite Lens | 17
  comfilcon A | 50
  No preference | 33

21. Secondary Outcome: Subjective Lens Preference -Overall Vision Preference
Description: Patient subjective preference: Phenacite test lens, comfilcon A or No Preference
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 30
percentage of participants
  Phenacite | 27
  comfilcon A | 56
  No Preference | 17

22. Secondary Outcome: Subjective Lens Preference - Comfort
Description: Patient subjective preference: Phenacite test lens, comfilcon A or No Preference
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 30
percentage of participants
  Phenacite | 43
  comfilcon A | 40
  No preference | 17

23. Secondary Outcome: Subjective Overall Lens Preference
Description: Patient subjective overall preference: Phenacite test lens, comfilcon A or No Preference
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 30
percentage of participants
  Phenacite | 33
  comfilcon A | 57
  No preference | 10

ADVERSE EVENTS:
Time Frame: From dispense up to one week on each study lens, a total of 2 weeks.
Arm/Group | Phenacite Contact Lens | Comfilcon A Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No